CLINICAL TRIAL: NCT04456764
Title: Real-time Intervention to Reduce Fatigue Among Emergency Medical Services Workers: A Cluster-randomized Trial
Brief Title: The Sleep and Teamwork in EMS Study
Acronym: SaFTiE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Performance period ended
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel Patterson, PhD, NRP, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19040354; R01OH011502 (NIH)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Fatigue; Sleep
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SaFTiE (Experimental): The SaFTiE intervention includes: [a] real-time text-message assessments of fatigue and sleep during and between scheduled shift work; [b] tailored text-message alerts that promote adopting evidence based strategies for mitigating fatigue when high levels of fatigue or sleepiness are reported; [c] a mobile app that delivers goal setting, summary data of sleep/fatigue indicators from all study participants, and video interviews of EMS clinicians focused on sleep and fatigue.
  Interventions: Behavioral: SaFTiE
- Attention Placebo Control (Placebo Comparator): The attention placebo control includes: [a] real-time text-message assessments of teamwork during and between scheduled shift work; [b] text-message alerts that promote techniques for mitigating poor teamwork when episodes of poor teamwork are reported; [c] a mobile app that delivers goal setting, summary data of teamwork indicators from all study participants, and video interviews of EMS clinicians focused on teamwork.
  Interventions: Behavioral: Attention Placebo Control

INTERVENTIONS:
Behavioral: SaFTiE — A multi-modal fatigue risk management program.
  Arms: SaFTiE
Behavioral: Attention Placebo Control — A multi-modal teamwork assessment program.
  Other Names: Teamwork
  Arms: Attention Placebo Control

SUMMARY:
More than half of Emergency Medical Services (EMS) workers report work-related mental and physical fatigue. Odds of injury among fatigued EMS workers are nearly double that of non-fatigued workers. There is a compelling need to reduce fatigue among EMS workers, yet few EMS organizations have a formal fatigue management program and many may not be cost-effective or evidence-based. This trial addresses national goals of the National Occupational Research Agenda (NORA) and tests a novel approach to fatigue risk management that is easily scalable to large workforces and low-cost for employers of shift workers.

DETAILED DESCRIPTION:
The investigators will test an enhanced version of our SleepTrackTXT pilot intervention - Sleep and Fatigue Treatment in EMS (SaFTiE) - in a two-arm parallel cluster-randomized design of EMS agencies. Our unit of randomization will be the EMS agency, with the intervention deployed as a Fatigue Risk Management Program that can be integrated into an agency's existing program. During the active intervention phase, the investigators will use SaFTiE and an attention placebo control (APC) group to test the specific effect of our multi-component intervention on EMS worker fatigue and sleep health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Live in United States (including Hawaii and Alaska)
* Licensed / certified EMS clinician
* Currently work in shifts
* Do at least one clinical shift per week
* Own a smartphone
* Willing to answer monthly surveys and daily text-messages,

Exclusion Criteria:

* Exclude EMS personnel who are primarily administrative with non-clinical duties
* Are restricted from using personal smartphone during periods of work
* Do not own a smartphone capable of running the study mobile app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. Daniel Patterson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will work with NIOSH/CDC and share de-identified research data via a NIOSH/CDC or NIH managed repository if requested. The study team will develop a process to receive requests from outside the study team for de-identified datasets should there be no NIOSH/CDC supported data repository.
Supporting Information: Study Protocol
Time Frame: Following publication of the primary study papers with primary and secondary outcomes reported.
Access Criteria: The study team will develop a process to receive requests from outside the study team for de-identified datasets should there be no NIOSH/CDC supported data repository.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: EMS Agencies
Period: Overall Study
Arm/Group | SaFTiE | Attention Placebo Control
Started | 385; 54 EMS Agencies | 323; 54 EMS Agencies
Completed | 319; 47 EMS Agencies | 272; 44 EMS Agencies
Not Completed | 66; 7 EMS Agencies | 51; 10 EMS Agencies

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SaFTiE | Attention Placebo Control | Total
Number analyzed (Participants) | 385 | 323 | 708
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Among participants who provided information on Age
  years
    number analyzed (Participants) | 371 | 318 | 689
    (all) | 37.7 (10.6) | 35.3 (9.8) | 36.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Among participants who provided information on sex
  Participants
    number analyzed (Participants) | 370 | 317 | 687
    Female | 138 | 105 | 243
    Male | 232 | 212 | 444
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Among participants who provided information on Ethnicity
  Participants
    number analyzed (Participants) | 368 | 315 | 683
    Hispanic or Latino | 24 | 12 | 36
    Not Hispanic or Latino | 339 | 298 | 637
    Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Among participants who provided information on Race
  Participants
    number analyzed (Participants) | 371 | 318 | 689
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 5 | 1 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 4 | 12
    White | 339 | 301 | 640
    More than one race | 14 | 8 | 22
    Unknown or Not Reported | 4 | 4 | 8
Chalder Fatigue Questionnaire (CFQ) [Mean (Standard Deviation); unit: units on a scale] — Population: Among participants who provided information on Chalder Fatigue Questionnaire (CFQ)
  units on a scale
    number analyzed (Participants) | 369 | 316 | 685
    (all) | 5.3 (2.9) | 5.2 (3.1) | 5.3 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Fatigue
Description: A response of 4 or greater on the Chalder Fatigue Questionnaire (CFQ) [minimum score=0, maximum score=11, and scores >=4 indicate mental and physical fatigue]
Time Frame: At baseline, 3 months, and 6 months
Population: Among participants who provided survey data
Measure: Count of Participants; unit: Participants
Arm/Group | SaFTiE | Attention Placebo Control
Number analyzed (Participants) | 369 | 316
Participants
  Baseline | 260 | 219
  3 months: number analyzed (Participants) | 263 | 219
  3 months | 172 | 122
  6 months: number analyzed (Participants) | 240 | 206
  6 months | 144 | 107
Statistical Analysis 1: Comparison: SaFTiE vs Attention Placebo Control; Test type: Superiority; p = 0.55, Mixed Models Analysis — Test for group by time interaction; Adjusted for clustering

2. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI measures sleep quality using a survey instrument with scores ranging from 0 to 21. Higher scores indicate poorer sleep quality.
Time Frame: Baseline, 3 months, and 6 months
Population: Among participants who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SaFTiE | Attention Placebo Control
Number analyzed (Participants) | 369 | 316
score on a scale
  Baseline | 9.0 (3.5) | 8.8 (3.8)
  3 months: number analyzed (Participants) | 263 | 219
  3 months | 7.9 (3.6) | 7.9 (4.0)
  6 months: number analyzed (Participants) | 240 | 206
  6 months | 7.4 (3.6) | 7.5 (3.7)
Statistical Analysis 1: Comparison: SaFTiE vs Attention Placebo Control; Test type: Superiority; p = 0.12, Mixed Models Analysis — group x time interaction; random agency and a random participant effect

3. Secondary Outcome: Poor Sleep Quality
Description: A response of 6 or greater on the Pittsburgh Sleep Quality Index (PSQI) [minimum score=0, maximum score=21, and scores >=6 indicate poor sleep quality]
Time Frame: At 6 months
Population: Among participants who reported poor sleep at baseline and had survey data at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SaFTiE | Attention Placebo Control
Number analyzed (Participants) | 240 | 206
Participants | 188 | 177
Statistical Analysis 1: Comparison: SaFTiE vs Attention Placebo Control; Test type: Superiority; p = 0.0986, Mixed Models Analysis; Adjusted for clustering

4. Secondary Outcome: Inter-Shift Recovery Measure
Description: This is the Inter-Shift Recovery sub-scale of the Occupational Fatigue Exhaustion Recovery (OFER) questionnaire. Individual item responses are coded 0 to 6 and summed, divided by 30, then multiplied by 100 to produce a composite sub-scale score ranging from 0 to 100. Higher scores on the inter-shift sub-scale signify greater/improved ability to recover between shifts. The OFER has no minimum thresholds to define clinically meaningful change in fatigue or recovery.
Time Frame: At baseline, 3 months, and 6 months
Population: Among participants who answered the OFER survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SaFTiE | Attention Placebo Control
Number analyzed (Participants) | 369 | 316
score on a scale
  Baseline | 51.4 (25.6) | 55.0 (25.1)
  At 3 months: number analyzed (Participants) | 263 | 219
  At 3 months | 52.0 (25.2) | 57.1 (24.7)
  At 6 months: number analyzed (Participants) | 240 | 206
  At 6 months | 52.3 (24.9) | 55.7 (25.1)
Statistical Analysis 1: Comparison: SaFTiE vs Attention Placebo Control; Test type: Superiority; p = 0.51, Mixed Models Analysis — Group by time interaction; Adjusted for clustering

5. Secondary Outcome: Acute Fatigue Measure
Description: This is the Acute Fatigue sub-scale of the Occupational Fatigue Exhaustion Recovery (OFER) questionnaire. Individual item responses are coded 0 to 6 and summed, divided by 30, then multiplied by 100 to produce a composite sub-scale score ranging from 0 to 100. Higher scores on the acute fatigue sub-scale (e.g., 50-100) signify moderate to high acute fatigue. The OFER has no minimum thresholds to define clinically meaningful change in fatigue or recovery.
Time Frame: Baseline, 3 months, and 6 months
Population: Among participants who answered the OFER survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SaFTiE | Attention Placebo Control
Number analyzed (Participants) | 369 | 316
score on a scale
  Baseline | 59.8 (23.7) | 57.6 (25.1)
  3 months: number analyzed (Participants) | 263 | 219
  3 months | 58.7 (24.7) | 52.8 (25.1)
  6 months: number analyzed (Participants) | 240 | 206
  6 months | 58.6 (23.4) | 56.1 (24.0)
Statistical Analysis 1: Comparison: SaFTiE vs Attention Placebo Control; Test type: Superiority; p = 0.04, Mixed Models Analysis — Group by time interaction; Adjusted for clustering

6. Secondary Outcome: Chronic Fatigue Measure
Description: This is the Chronic Fatigue sub-scale of the Occupational Fatigue Exhaustion Recovery (OFER) questionnaire. Individual item responses are coded 0 to 6 and summed, divided by 30, then multiplied by 100 to produce a composite sub-scale score ranging from 0 to 100. Higher scores on the chronic fatigue sub-scales (e.g., 50-100) signify moderate to high chronic fatigue. The OFER has no minimum thresholds to define clinically meaningful change in fatigue or recovery.
Time Frame: Baseline, 3 months, 6 months
Population: Among participants who answered the OFER survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SaFTiE | Attention Placebo Control
Number analyzed (Participants) | 369 | 316
score on a scale
  Baseline | 35.8 (25.0) | 32.7 (24.4)
  3 months: number analyzed (Participants) | 263 | 219
  3 months | 38.9 (26.6) | 33.9 (25.3)
  6 months: number analyzed (Participants) | 240 | 206
  6 months | 38.8 (26.5) | 37.2 (26.8)
Statistical Analysis 1: Comparison: SaFTiE vs Attention Placebo Control; Test type: Superiority; p = 0.02, Mixed Models Analysis — Group by time interaction; Adjusted for clustering

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for this study.
Arm/Group | SaFTiE | Attention Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination prior to reaching goal enrollment leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04456764/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT04456764/ICF_000.pdf